CLINICAL TRIAL: NCT01546025
Title: Brief Alcohol Intervention for School-to-Work Transitions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Suzanne M. Colby, Associate Professor, Research, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA016000 (NIH); R01AA016000 (NIH)
Record Dates: First submitted 2012-02-20; First posted 2012-03-07 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Binge Drinking
MeSH Terms: conditions — Binge Drinking | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Relaxation training (REL) (Placebo Comparator): This was a 1-hr behavioral counseling session designed to control for nonspecific therapeutic effects by providing equivalent levels of attention from and rapport with a counselor. It began with an introduction and rapport building. The counselor asked about the participant's daily stress level and strategies used to cope. Experience with meditation and relaxation were explored. The counselor presented a rationale for the use of REL for alcohol reduction, namely: the transition to adulthood can be stressful, and stress can lead to increased alcohol use; meditation and relaxation can reduce stress and thereby prevent excessive alcohol use. Didactic information about mental and physical stress and coping was provided. Two strategies were practiced: a simple, guided breathing meditation and a full-body progressive muscle relaxation. The session concluded with a review of the participant's experiences during the 2 exercises and a recommendation to practice the techniques regularly.
  Interventions: Behavioral: Relaxation training
- Brief Motivational Intervention (BMI) (Active Comparator): This is a 1-hr motivational intervention session. The counselor built rapport while eliciting information about the participant's drinking, discussing current experiences, goals and plans in different domains (education, work, financial independence, social transitions, relationships). The counselor explored how drinking fit into the participant's life and explored risk and protective factors. The session involved: Assessing motivation; Enhancing motivation; Personalized feedback; Envisioning the future with/without change; Counselor summary; and Optional personalized change plan. Participant strengths, protective factors, and autonomy/ability to make changes were elicited and supported. Counselors used MI principles and techniques, including using open-ended questions, reflective listening, eliciting change talk, and supporting self-efficacy statements.
  Interventions: Behavioral: Brief Motivational Counseling

INTERVENTIONS:
Behavioral: Brief Motivational Counseling — One hour session of brief motivational counseling focused on reduction of heavy drinking.
  Other Names: Brief Motivational Intervention; BMI
  Arms: Brief Motivational Intervention (BMI)
Behavioral: Relaxation training — One hour training in relaxation techniques
  Other Names: REL
  Arms: Relaxation training (REL)

SUMMARY:
This is a 2-year research project to test the efficacy of brief motivational intervention for reducing heavy alcohol use in young adults transitioning out of high school. Participation occurs within 3 months prior to graduation or within 1 year following graduation or dropout from high school. Heavy drinkers ages 17-20 will be randomly assigned to receive one session of BMI or one session of relaxation training. All participants complete identical assessments at baseline and immediately post-intervention (during session 1). Participants also complete in-person 6-week and 3-month follow up assessments to evaluate intervention effects. Study aims involve: a) testing the comparative efficacy of BMI; b) identifying moderators (person-level predictors) of intervention response; and c) identifying mediators (mechanisms) of intervention effects, that is, how BMI exerts its effect on outcomes.

DETAILED DESCRIPTION:
This study tested the efficacy of a single session of BMI for reducing heavy drinking and related adverse consequences among underage young adult drinkers not attending a 4-year college or university. We designed the intervention to be delivered proximal to the transition out of high school (with or without graduation), because such periods of transition and discontinuity in the life course present opportunities to positively alter developmental paths (Masten et al., 2009). Thus, interventions timed to co-occur with naturalistic transition points may have great potential for decreasing drinking trajectories or preventing harmful escalations in trajectories going forward. To increase the applicability of our findings to the heterogeneous population of community-dwelling young adults, our recruitment targeted a purposefully inclusive "non-4-year-college" population. We hypothesized that, compared to a time and attention-matched control condition (i.e., relaxation training [REL]), BMI would result in significantly reduced heavy drinking and reduced adverse consequences of alcohol use at 6-week and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* high school students anticipating graduation within 3 months, drop outs or graduates
* males must report at least one day drinking 5 or more standard drinks in past month
* females must report at least one day drinking 4 or more standard drinks in past month

Exclusion Criteria:

* plans to enroll at traditional 4-year college within 12 months
* plans to enter military within next 12 months
* plans to move more than 1 hour from current location in within 12 months

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

REFERENCES:
- [Result] Colby SM, Orchowski L, Magill M, Murphy JG, Brazil LA, Apodaca TR, Kahler CW, Barnett NP. Brief Motivational Intervention for Underage Young Adult Drinkers: Results from a Randomized Clinical Trial. Alcohol Clin Exp Res. 2018 Jul;42(7):1342-1351. doi: 10.1111/acer.13770. Epub 2018 Jun 6. PMID 29750362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was promoted via posted flyers in the community; advertisements on buses, websites, and in newspapers; and recruitment events at high schools, community colleges, vocational/technical programs, social service agencies, and GED classes. Research staff described the study to groups/classes or at information booths set up in a lobby or cafeteria. Data collection took place in Rhode Island and Southeastern Massachusetts from June 2010 to October 2011.
Pre-assignment Details: 168 were consented and enrolled. One person was determined to be ineligible because they were simultaneously participating in another alcohol intervention research study simultaneously. That were person was withdrawn from the study, resulting in a sample of 167 participants.
Period: Overall Study
Arm/Group | Relaxation Training | Brief Motivational Counseling
Started | 84 (randomly assigned to Relaxation Training (REL)) | 83 (randomly assigned to Brief Motivational Intervention (BMI))
Completed Treatment | 84 | 83
6-week Follow up | 82 | 80
3-month Follow up | 81 | 80
Completed (Analysis sample: completed at least one follow up) | 84 | 82
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Relaxation Training: Relaxation training (REL): One hour training in relaxation techniques REL was designed to control for nonspecific therapeutic effects by providing equivalent levels of attention from and rapport with a counselor. REL began with an introduction to the intervention and general rapport building. The counselor asked about the participant's typical experiences with daily stress, and reviewed various strategies the participant had used to cope with stress. Past experiences with meditation and relaxation were explored. To promote positive treatment expectancies, the counselor presented a rationale for the use of REL for alcohol reduction. Participants were told: (i) the transition to adulthood can be stressful, and stress can lead to increased alcohol use; and (ii) alternative approaches to coping with stress, such as meditation and relaxation techniques, can reduce stress and thereby prevent excessive alcohol use. For the remainder of the session, 2 strategies for coping with stress were introduced and practiced: the first was a simple, guided breathing meditation; and the second was a full-body progressive muscle relaxation. Both exercises were scripted and read aloud by the counselor as the participant followed the counselor instructions. The session concluded with a review of the participant's experiences during the 2 exercises and a counselor recommendation to practice the techniques regularly.
- Brief Motivational Counseling: Brief Motivational Intervention (BMI) Counseling: One hour session of BMI focused on reduction of heavy drinking. The counselor built rapport while eliciting information about the developmental context of the participant's drinking behavior, discussing current experiences, goals, and plans for the next several years in different domains (education/training, work, financial independence, social transitions, romantic relationships). The counselor explored how alcohol and drinking fit into the participant's life, and how the participant expected their drinking to change into adulthood. Assessing motivation involved exploring the positive and negative aspects of drinking for participants. Enhancing motivation consisted of providing a personalized feedback report including normative feedback, and personalized risk factors and other elements like time and money allocation. Participants were asked to envision themselves in the future if they decided to make a change, and again if they decided not to change. The counselor drew upon participants' goals (e.g., social, recreational, occupational, financial) to highlight discrepancies between drinking behavior and proximal life goals. The participant identified goals for change related to drinking. The BMI reviewed strategies for reducing heavy drinking. Participant strengths, protective factors, and autonomy/ability to make changes were elicited and supported. Throughout the session, counselors used MI principles and techniques.
- Total: Total of all reporting groups
Arm/Group | Relaxation Training | Brief Motivational Counseling | Total
Number analyzed (Participants) | 84 | 83 | 167
Age, Customized [Count of Participants; unit: Participants]
  age 17 | 22 | 24 | 46
  age 18 | 30 | 29 | 59
  age 19 | 24 | 19 | 43
  age 20 | 8 | 11 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 48 | 49 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 8 | 10 | 18
  Non-Hispanic White | 51 | 48 | 99
  Non-Hispanic Black/African American | 7 | 9 | 16
  American Indian/Native American | 0 | 1 | 1
  Asian/Pacific Islander | 6 | 1 | 7
  More than 1 race | 12 | 11 | 23
  missing | 0 | 3 | 3
Avg Number of Standard Drinks per week [Mean (Standard Deviation); unit: standard drinks per week] — This is a calculation of estimated average drinks consumed per week at baseline, using daily data derived from the timeline follow back interview
  standard drinks per week | 12.14 (8.85) | 14.85 (14.41) | 13.49 (12.36)

OUTCOME MEASURES:

1. Primary Outcome: Timeline Follow Back Assessing Number of Standard Drinks
Description: This is a calculation of the number of standard alcohol drinks consumed per week, based on data collected via the timeline follow back interview
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: standard drinks/week
Arm/Group | Relaxation Training | Brief Motivational Counseling
Number analyzed (Participants) | 81 | 80
standard drinks/week | 8.93 (10.00) | 5.56 (5.91)

2. Secondary Outcome: Brief Young Adult Alcohol Consequences Questionnaire
Description: Measure of problem severity in young adult drinkers. Respondents indicated on the Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ; Kahler et al., 2005) whether they had experienced each of 24 adverse alcohol-related consequences in the prior 6 weeks; items are summed for a total score (Cronbach's α = 0.81 at BL), with a minimum score of 0 and a maximum score of 24. Higher scores indicate worse outcome.
Time Frame: 6 week and 3 month follow ups
Population: This measure is analyzed among participants who reported any alcohol use in the assessment window.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Training | Brief Motivational Counseling
Number analyzed (Participants) | 70 | 71
units on a scale
  Brief Young Adult Alcohol Consequences Questionnaire 6 weeks | 6.43 (0.50) | 5.47 (0.49)
  Brief Young Adult Alcohol Consequences Questionnaire 3 months | 6.01 (0.52) | 4.85 (0.51)

3. Secondary Outcome: Help Seeking
Description: Count of participants reporting receiving any type of counseling for alcohol in the prior 6 weeks
Time Frame: 6 week and 3 month follow ups
Population: Participants in each group with data on this variable at 6 week follow up and 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Relaxation Training (REL) | Brief Motivational Intervention (BMI)
Number analyzed (Participants) | 81 | 80
Participants
  Number reporting alcohol counseling, 6 week follow up | 10 | 9
  Number reporting alcohol counseling, 3 month follow up | 6 | 8

4. Secondary Outcome: Drinking Reduction Strategies
Description: Total score on the Strategies to Limit Drinking 31-item scale. Likert response for each item ranges from 1 = never to 5 = always; range = 31 to 155; higher scores indicate better outcomes: higher scores reflect greater frequency of using various strategies to deliberately limit one's drinking over the past 6 weeks
Time Frame: 6 week and 3 month follow ups
Population: Participants in each group with data on this variable at 6 week and 3 month follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Training (REL) | Brief Motivational Intervention (BMI)
Number analyzed (Participants) | 82 | 81
units on a scale
  Drinking reduction score, 6 week follow up: number analyzed (Participants) | 82 | 80
  Drinking reduction score, 6 week follow up | 94.6 (27.7) | 99.6 (27.4)
  Drinking reduction score, 3 month follow up: number analyzed (Participants) | 81 | 80
  Drinking reduction score, 3 month follow up | 89.9 (29.8) | 98.6 (31.1)

5. Secondary Outcome: Employment Outcomes
Description: Mean score on the "Your Workplace" questionnaire: Negative Effects on Work Performance subscale.
  Range = 0 to 5. Response options for each item on the subscale are 0 = never; 1 = once or twice, 2 = about once every 2 weeks, 3 = about once a week, 4 = 2-4 times a week, 5 = about daily.
  Higher scores indicate worse outcomes: Higher scores reflect more frequent negative effects of alcohol use on work performance in the past 6 weeks.
Time Frame: 6 week and 3 month follow ups
Population: This includes all participants in each group at 6 week and at 3 month follow up who reported engaging in paid employment in the prior 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Training (REL) | Brief Motivational Intervention (BMI)
Number analyzed (Participants) | 59 | 52
units on a scale
  Negative alcohol effects at work, 6 week follow up | 0.16 (0.44) | 0.13 (0.31)
  Negative alcohol effects at work, 3 month follow up | 0.14 (0.51) | 0.12 (0.28)

6. Secondary Outcome: Satisfaction With Life
Description: This is a mean score on the Satisfaction With Life Scale (SWLS), a 5-item instrument designed to measure global cognitive judgments of life satisfaction, using a 7-point Likert scale (1=strongly disagree to 7=strongly agree), with higher scores indicating better outcomes, i.e., higher scores indicate greater life satisfaction at the time of assessment. Range = 1 to 7.
Time Frame: 6 week and 3 month follow ups
Population: Participants in each group with valid data on this scale at 6 week or 3 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Relaxation Training (REL) | Brief Motivational Intervention (BMI)
Number analyzed (Participants) | 82 | 80
units on a scale
  General life satisfaction, 6 week follow up | 4.80 (1.43) | 4.72 (1.25)
  General life satisfaction, 3 monnth follow up: number analyzed (Participants) | 81 | 80
  General life satisfaction, 3 monnth follow up | 4.96 (1.41) | 4.95 (1.20)

7. Secondary Outcome: Adolescent Reinforcement Survey Schedule (ARSS)
Description: The ARSS contains a list of 45 rewarding activities. Participants rate the frequency with which they participate in each activity WITH and then WITHOUT alcohol/drug use, and then rate their enjoyment of each activity WITH and WITHOUT alcohol/drug use. The outcome measure represents the percentage of reinforcement participants get (i.e., the cross product of frequency X enjoyment) from activities involving alcohol/drug use divided by the total reinforcement they get from all activities with or without alcohol/drug use. Range = 0 to 100; higher scores indicate worse outcomes, i.e., higher scores reflect a greater percentage of enjoyable activities involving alcohol and/or use.
Time Frame: 6 week and 3 month follow ups
Population: Participants in each group with valid data on this variable at 6 week or 3 month follow up.
Measure: Mean (Standard Deviation); unit: percentage of enjoyment due to alcohol
Arm/Group | Relaxation Training (REL) | Brief Motivational Intervention (BMI)
Number analyzed (Participants) | 82 | 80
percentage of enjoyment due to alcohol
  Enjoyment attributed to alcohol, 6 week follow up | 33.7 (18.9) | 32.7 (19.3)
  Enjoyment attributed to alcohol, 3 month follow up: number analyzed (Participants) | 82 | 79
  Enjoyment attributed to alcohol, 3 month follow up | 29.4 (21.0) | 30.0 (18.7)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Any adverse events reports at study contacts were to be recorded in study record.
Arm/Group | Relaxation Training | Brief Motivational Counseling
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/83
Other Adverse Events (participants affected / at risk) | 0/84 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No